CLINICAL TRIAL: NCT07179250
Title: Effect of Breathing Training on Symptoms of Gastroesophageal Reflux Disease: A Parallel Randomized Controlled Trial
Brief Title: Effect of Breathing Training on Symptoms of Gastroesophageal Reflux Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCH-IRB-250618; CCH-IRB-250618 (Other Grant/Funding Number: Changhua Christian Hospital)
Record Dates: First submitted 2025-09-11; First posted 2025-09-17 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Incentive Spirometer; Diaphragmatic Breathing; Gastroesophageal Reflux Disease (GERD); Breath Exercise
Keywords: GERD; Gastroesophageal Reflux Disease; Acid Reflux; Diaphragmatic Breathing; Breathing Training; Incentive Spirometer; Volume-Oriented Incentive Spirometry; GERDQ; Gastroesophageal Reflux Disease Questionnaire; breath exercise
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial adopts a parallel assignment model with three arms: volume-oriented incentive spirometry (VIS), diaphragmatic breathing exercise (DBE), and usual care (control). Participants are randomized in a 1:1:1 ratio using a computer-generated sequence with allocation concealment through sealed opaque envelopes. The intervention period lasts 6 weeks, and assessments are performed at baseline and week 7. No crossover between groups is planned.
Who Masked: Outcomes Assessor
Masking Description: This study uses a single-blind design. Outcome assessors analyzing GERDQ questionnaires, high-resolution manometry, and 24-hour pH-impedance data are blinded to group assignments, while participants, care providers, and investigators are aware of interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Volume-Oriented Incentive Spirometry (VIS) (Experimental): Participants in this group will perform diaphragmatic breathing exercises twice daily for 6 weeks using a volume-oriented incentive spirometer, in addition to usual care. Assessments will be conducted at baseline and at the end of week 7.
  Interventions: Device: Volume-Oriented Incentive Spirometer
- Diaphragmatic Breathing Exercises (DBE) (Experimental): In this group will perform standard diaphragmatic breathing exercises twice daily for 6 weeks, in addition to usual care. Assessments will be conducted at baseline and at the end of week 7.
  Interventions: Behavioral: Diaphragmatic Breathing Exercise (DBE)
- Usual Care (Control) (Placebo Comparator): Participants in this group will receive standard clinical management for gastroesophageal reflux disease without structured breathing training. Assessments will be conducted at baseline and at the end of week 7.
  Interventions: Behavioral: Usual Care and Education

INTERVENTIONS:
Device: Volume-Oriented Incentive Spirometer — Participants in the experimental group will perform volume-oriented incentive spirometry training twice daily (morning and evening) for 6 weeks. Each session consists of 10 deep inspirations using the spirometer, with the target volume initially set according to the participant's predicted maximum inspiratory capacity and increased by approximately 5% each week starting from week 2. For each breath, participants inhale to reach the target volume, hold their breath for 3-5 seconds, and then exhale. A rest period of 30-60 seconds is allowed between maneuvers, and the pace is adjusted according to individual tolerance. Training is performed in a seated or semi-recumbent position.
  Arms: Volume-Oriented Incentive Spirometry (VIS)
Behavioral: Diaphragmatic Breathing Exercise (DBE) — Participants in the control group will perform diaphragmatic breathing exercises twice daily (morning and evening) for 6 weeks. During weeks 1-2, each session consists of 10 breaths per set; from week 3 to week 6, each session consists of 15 breaths per set. The exercise is performed without devices and includes the following sequence: slow inspiration through the nose with abdominal expansion, holding the breath for 5 seconds, followed by exhalation through the mouth with visible abdominal contraction. After each set, participants rest with natural breathing for 1-2 minutes to prevent hyperventilation or diaphragmatic fatigue. Training is conducted in a semi-recumbent position with both hands placed behind the head, focusing on abdominal movement control and breathing rhythm.
  Arms: Diaphragmatic Breathing Exercises (DBE)
Behavioral: Usual Care and Education — Participants in the control group will receive usual clinical care for gastroesophageal reflux disease (GERD) without structured breathing training. At study entry, participants are provided with standardized patient education regarding GERD and lifestyle modification strategies, along with an educational leaflet. No specific posture or breathing exercises are required during the study period.
  Arms: Usual Care (Control)

SUMMARY:
The goal of this clinical trial is to evaluate whether two types of breathing training can improve symptoms of gastroesophageal reflux disease (GERD) in adults.

The main research questions are:

* Do volume-oriented incentive spirometry (VIS) or diaphragmatic breathing exercise (DBE) improve GERD symptoms compared with usual care?
* Do these breathing exercises reduce the symptoms of GERD?
* Does volume-oriented incentive spirometry (VIS) produce greater improvement in GERD symptoms compared with DBE?
* Do these exercises increase the strength of the lower esophageal sphincter (LES)?

Researchers will compare VIS training, DBE training, and usual care to determine whether breathing training can serve as a safe and effective non-pharmacological treatment option for GERD.

Participants will:

* Be randomly assigned to VIS training, DBE training, or usual care
* Perform their assigned breathing training (if in the intervention group) twice daily for 6 weeks
* Attend study visits at baseline and at week 7 for questionnaires and esophageal function tests
* Keep a diary of their symptoms and breathing practice

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is a prevalent gastrointestinal disorder resulting from dysfunction of the lower esophageal sphincter (LES) and impaired anti-reflux barrier mechanisms. While proton pump inhibitors (PPIs) are effective in reducing gastric acid secretion, up to 30-40% of patients report persistent symptoms despite optimized medical therapy. Non-pharmacological interventions are therefore of growing clinical interest.

Diaphragmatic breathing exercise (DBE) targets abdominal breathing patterns to enhance diaphragmatic tone and coordination. This may improve the esophagogastric junction competence and reduce transient LES relaxations. Volume-oriented incentive spirometry (VIS), a device providing visual feedback during sustained deep inspiration, has been demonstrated to facilitate diaphragmatic recruitment and strengthen inspiratory effort. VIS has shown benefits in perioperative recovery, pulmonary rehabilitation, and post-COVID-19 recovery, but has not yet been systematically studied in GERD populations.

This randomized controlled trial adopts a parallel three-arm design, comparing VIS training, DBE training, and a usual care control group. Participants in the intervention arms will be instructed to perform their assigned breathing training twice daily for six weeks. Standardized protocols will be applied: VIS training will target 80-90% of predicted inspiratory capacity with 3-5 seconds of breath-hold at peak inspiration, while DBE will emphasize abdominal expansion and controlled diaphragmatic contraction.

Objective outcome measures include high-resolution manometry (HRM) to assess LES basal pressure and 24-hour pH-impedance monitoring to quantify esophageal acid exposure time (AET) and reflux episodes. GERD symptom severity will be evaluated using validated questionnaires (GERDQ). Assessments are scheduled at baseline and week 7 following the intervention.

The primary hypothesis is that both VIS and DBE will improve GERD symptoms compared with usual care, with VIS expected to demonstrate superior enhancement of diaphragmatic activation and LES pressure. Secondary outcomes will explore physiological changes in esophageal acid exposure, symptom-reflux association, and intervention feasibility.

This trial is expected to generate evidence supporting safe, low-cost, and accessible non-pharmacological strategies for GERD management, complementing or potentially reducing the need for long-term pharmacotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20 to 80 years
* Endoscopic finding of reflux esophagitis (LA grade A) with proton pump inhibitor (PPI) use > 2 months, or 24-hour pH monitoring showing acid exposure time (AET) > 6%, or endoscopic diagnosis of reflux esophagitis LA grade B or higher
* Willingness to comply with the full training and follow-up protocol

Exclusion Criteria:

* Pregnant or breastfeeding women
* History of anti-reflux surgery
* Severe cardiopulmonary dysfunction or respiratory disease
* Inability to perform the training exercises or attend follow-up visits

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in lower esophageal sphincter (LES) pressure | Baseline and Week 7
  LES pressure will be measured using high-resolution manometry (HRM). The mean resting pressure (mmHg) of the LES will be recorded and analyzed to evaluate changes from baseline to week 7 between groups

SECONDARY OUTCOMES:
Change in GERD symptom severity measured by GERDQ | Baseline and Week 7
  GERD-related symptoms will be assessed using the Gastroesophageal Reflux Disease Questionnaire (GERDQ), a validated 6-item self-reported instrument. The total score ranges from 0 to 18, with higher scores indicating more severe symptoms. Changes from baseline to week 7 will be compared between groups.
Change in the number of reflux episodes within 24 hours | Baseline and Week 7
  Ambulatory 24-hour pH-impedance monitoring will be used to quantify the total number of gastroesophageal reflux episodes. Differences between baseline and week 7 will be assessed across groups
Change in esophageal acid exposure time (AET) | Baseline and Week 7
  Esophageal acid exposure will be evaluated using 24-hour pH monitoring. AET is defined as the percentage of time with esophageal pH < 4.0 during the 24-hour monitoring period. Changes from baseline to week 7 will be compared
Change in the number of effective esophageal peristalsis events | Baseline and Week 7
  Esophageal motility will be assessed using high-resolution manometry (HRM). The number of effective peristaltic contractions within 24 hours will be recorded. Changes from baseline to week 7 will be analyzed between groups

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Ju Tu, MSN, NP, RN, Principal Investigator — Changhua Christian Hospital, Dept. of Gastroenterology

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared, including demographic characteristics, baseline clinical data, intervention adherence, and primary and secondary outcome measures (GERDQ scores, LES pressure, 24-hour pH-impedance results, and HRM parameters). No identifiable personal information will be included.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified individual participant data and supporting information (study protocol, SAP) will be available beginning 6 months after publication of the primary results. Data will remain available for 3 years after publication.
Access Criteria: Data will be available to qualified researchers for purposes of meta-analysis or secondary research related to gastroesophageal reflux disease. Requests should be submitted to the Principal Investigator by email. Access will be granted after review and approval of a reasonable research proposal, and a data use agreement may be required.